CLINICAL TRIAL: NCT07052383
Title: A Single-Arm, Open-Label Clinical Study to Evaluate the Safety and Efficacy of DIT309 Cell Injection in Subjects With Advanced Bone and Soft Tissue Sarcomas
Brief Title: Safety and Efficacy of DIT309 in Advanced Bone and Soft Tissue Sarcomas
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tcelltech Inc. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIT309T-IS001
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Osteosarcoma; Soft Tissue Sarcoma
Keywords: Advanced
MeSH Terms: conditions — Osteosarcoma; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation Cohort (Experimental): DIT309 were administered via intravenous reinfusion on Days 1 in a 28-day treatment cycle.
  Interventions: Biological: DIT309 cell injection

INTERVENTIONS:
Biological: DIT309 cell injection — 3+3 dose escalation design： Dose Level 1: 4.0×10^6/kg CAR+ T cells；Dose Level 2: 1.0×10^7/kg CAR+ T cells；Dose Level 3: 2.0×10^7/kg CAR+ T cells.

SUMMARY:
This is a open-Label, dose-escalation study to evaluate the safety, tolerability and antitumor activity of DIT309 in subjects with advanced bone and soft tissue sarcomas.The study also plan to explore the Maximum Tolerated Dose (MTD) and determine the Recommended Phase II Dose (RP2D) of the CAR-T cell therapy.

DETAILED DESCRIPTION:
Subjects will be enrolled to receive DIT309 via intravenous infusion. Patients will be administered DIT309 on Day 1 of each 28-day treatment cycle, followed by a 28-day observation period.

The study will include three escalating dose levels, utilizing a traditional 3+3 dose escalation design. Each dose level will enroll 3 to 6 patients. Dose-limiting toxicities (DLTs) will be assessed during the first treatment cycle to evaluate the safety and tolerability of DIT309.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the clinical trial; is fully informed about the study and has signed the informed consent form (ICF); is willing and able to comply with all study procedures.
2. Male or female patients aged ≥8 weeks.
3. Histologically confirmed diagnosis of advanced bone and soft tissue sarcoma, who have failed or are intolerant to prior standard therapies.
4. At least one measurable lesion as defined by RECIST version 1.1.
5. B7-H3-positive tumor confirmed by pathological testing, with B7-H3 positivity defined as ≥20% B7-H3-positive tumor cells in non-necrotic tumor tissue.
6. ECOG performance status of 0-1 within 24 hours prior to leukapheresis and prior to lymphodepletion.
7. Life expectancy of more than 6 months.
8. Adequate venous access for leukapheresis, with no contraindications for the procedure.
9. Laboratory parameters must meet the following criteria:

   1. Hematologic function: WBC ≥ 3.0 × 10⁹/L; Hemoglobin ≥ 8.0 g/dL; ANC ≥ 1.5 × 10⁹/L; Platelets ≥ 75.0 × 10⁹/L
   2. Renal function: Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
   3. Hepatic function: ALT and AST ≤ 2.5 × ULN (≤ 5.0 × ULN for subjects with liver metastasis)
   4. Total bilirubin ≤ 2.0 × ULN (excluding patients with Gilbert's syndrome, defined as persistent or recurrent unconjugated hyperbilirubinemia without evidence of hemolysis or hepatic pathology)
   5. Coagulation: Without anticoagulation therapy, PT, APTT, or INR ≤ 1.5 × ULN
   6. Negative pregnancy test for female subjects of childbearing potential
10. Subjects of childbearing potential must agree to use effective contraception from the date of signing the informed consent through 6 months after the last infusion.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Viral infections:

   1. Positive serology for HIV antibodies or syphilis
   2. Positive HBsAg or HBcAb with HBV DNA above the lower limit of detection in peripheral blood
   3. Positive HCV antibody with detectable HCV RNA in peripheral blood
3. Medical history and comorbidities:

   1. Known hypersensitivity to DIT309 cells or any component of the investigational products (including fludarabine, cyclophosphamide, or trastuzumab), or history of severe allergic reactions
   2. Known active autoimmune diseases (e.g., Crohn's disease, systemic lupus erythematosus); subjects with vitiligo or childhood asthma in complete remission and not requiring treatment in adulthood may be eligible; subjects requiring medical intervention such as bronchodilators for asthma are not eligible
   3. Currently receiving systemic immunosuppressive therapy or anticipated need for long-term immunosuppression during the study (topical, inhaled, or intranasal corticosteroids used intermittently are allowed)
   4. Prior exposure to any gene-modified T cell therapy (e.g., CAR-T or TCR-T) or any form of gene therapy*
   5. History of uncontrolled neurological or psychiatric disorders that may increase the risk of participation or interfere with study results in the investigator's opinion, including but not limited to epilepsy, dementia, or major depression
   6. Untreated or symptomatic CNS or leptomeningeal metastases
   7. Unresolved toxicities from prior treatment that have not recovered to Grade ≤1 per CTCAE v5.0 (except for toxicities deemed not to pose safety risk by the investigator, such as alopecia, Grade 2 peripheral neuropathy, or hypothyroidism managed with replacement therapy)
   8. History of other primary solid malignancies
   9. Major surgery or significant trauma within 1 month prior to leukapheresis
   10. Any serious or uncontrolled comorbidity that, in the investigator's opinion, may increase risks associated with study participation or investigational drug administration, including but not limited to: cardiovascular or cerebrovascular disease, renal insufficiency, pulmonary embolism, coagulation disorders requiring long-term anticoagulation, active or uncontrolled infections requiring systemic treatment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Safety：Incidence of Dose Limiting Toxicity (DLT) | 28 days after the first DIT309 infusion.
  Type, incidence, and severity of dose limiting toxicities (DLTs) within 28 days after the first DIT309 infusion.
Safety：Incidence and severity of adverse events (AEs) | 1year post CAR-T cells infusion.
  To evaluate the possible adverse events after DIT309 infusion, including the incidence, and severity of AEs.
The maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of DIT309. | From first dose of DIT309 until the end of Dose Limiting Toxicity (DLT) observation period (typically 28 days post-infusion for each dose cohort).
  The maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of DIT309.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year post CAR-T cells infusion.
  To evaluate the time from the start of DIT309 therapy to disease progression (according to RICIST1.1 criteria) or death from any cause, whichever occurs first.
  The proportion of progression-free subjects from the beginning of DIT309 therapy to a fixed time point (6 months) after treatment (6-Mon PFS) will also be evaluated.
Disease Control Rate (DCR) | 1 year post CAR-T cells infusion.
  To evaluate the proportion of subjects who achieved CR/PR/SD in the best overall response according to RICIST1.1 criteria.
Duration of disease control (DDC) | 1 year post CAR-T cells infusion.
  To evaluate the time from the first evaluation of tumor as CR, PR or SD to the first evaluation of PD or death from any cause.
Objective response rate (ORR) | 1 year post CAR-T cells infusion.
  To evaluate the proportion of subjects who achieved CR/PR in the best response condition according to RICIST1.1 criteria.
Time to Remission (TTR) | 1 year post CAR-T cells infusion.
  To evaluate the time from the start of treatment to the first remission (CR/PR).
Duration of Response (DOR) | 1 year post CAR-T cells infusion.
  DOR after DIT309 infusion, defined as the time from the first evaluation of the tumor as CR or PR to the first evaluation of PD or death from any cause.

OTHER OUTCOMES:
The immunogenicity of DIT309 | Up to 12 months
  Drug antibody (ADA) positive rate after infusion of DIT309 cells.
The positive rate of replication competent lentivirus tests | Up to 15 years.
  Detect replication competent lentivirus (RCL)
Peak Concentration (Cmax) of DIT309 CAR gene. | Up to 12 months
  Peak Concentration (Cmax) of DIT309 CAR gene.
Area under the concentration versus time curve (AUC) of DIT309 CAR-T cells | Area under the concentration versus time curve (AUC) of DIT309 CAR-T cells.
  Up to 12 months.
Peak concentration of cytokines | Up to 12 months
  Peak concentration of IL-2, IL-4，IL-6, IL-8，IL-10，IFN-γ， TNF-a

CONTACTS AND LOCATIONS:
Overall Officials: Gangxiong Huang, MD, Study Chair — Tcelltech Inc.
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No